CLINICAL TRIAL: NCT05564065
Title: Comparison of Intra-articular Steroid Injection and Radiofrequency Thermocoagulation of the Sensory Branches of the Femoral and Obdurator Nerves in Coxarthrosis Patients
Brief Title: Comparison of Intra-articular Steroid Injection and Radiofrequency Thermocoagulation in Coxarthrosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Halil Cetingok, Assistant professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/123
Record Dates: First submitted 2022-09-30; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Pain Hip Burning

STUDY DESIGN:
Intervention Model Description: Two groups: 1. intraarticular steroid injection of hip joint; 2. Radiofrequency thermocoagulation of femoral and obturator nerve terminal sensory branches of hip joint
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency thermocoagulation of sensory branches of hip joint (Active Comparator): There are two main nerves that carry the pain sensation of the hip joint. These nerves are the femoral and obturator nerves. The sensory branches of these nerves going to the hip joint will be detected with a radiofrequency device under fluoroscopy and percutaneous ablation will be performed.
  Interventions: Procedure: Radiofrequency thermocoagulation of sensory branches of hip joint
- Intraarticular steroid injection of hip joint (Active Comparator): Fluoroscopy guided percutaneous intra articular steroid injection of hip joint will be performed
  Interventions: Procedure: Intraarticular steroid injection of hip joint

INTERVENTIONS:
Procedure: Radiofrequency thermocoagulation of sensory branches of hip joint — There are two main nerves that carry the pain sensation of the hip joint. These nerves are the femoral and obturator nerves. The sensory branches of these nerves going to the hip joint will be detected with a radiofrequency device under fluoroscopy and percutaneous ablation will be performed.
  Arms: Radiofrequency thermocoagulation of sensory branches of hip joint
Procedure: Intraarticular steroid injection of hip joint — Fluoroscopy guided percutaneous intra articular steroid injection of hip joint will be performed
  Arms: Intraarticular steroid injection of hip joint

SUMMARY:
The investigators aimed that the Comparison of effectiveness of the intra-articular steroid injection and radiofrequency thermocoagulation of the sensory branches of the femoral and obdurator nerves in coxarthrosis patients

DETAILED DESCRIPTION:
Osteoarthirtis is a deficency of articular cartilge which is caused by genetic, metabolic and biochemical factors. This is a pathologic period with cartilage, bone and sinovium destruction.

Pharmacological treatments and/or phsiycal medicine may not be enough to reduce pain in patients with chronic pain of osteoarthiritis. Intraarticular steroid injection is the most common used intervention method in analgesia of hip osteoarthirtis. Thus; cartilage inflammation can be decelerated and osteophyte formation can be prevented. On the other hand; because of less vascularity of hip joint, frequent steroid injections may cause aseptic necrosis.

In past decades, treatment to pain of hip joint pain caused by ostheoarthrits, radiofrequency ablation treatment is used to sensory nerves which cause pain. Especially, it can be a solution in patients who do not want to undergo a surgery.

Patients diagnosed with coxarthrosis will be randomly divided into two groups. One group will receive intra-articular steroid injection and the other group will receive radiofrequency thermocoagulation to the hip sensory nerve branches (femoral and obdurator). It was planned to compare the vas scores of the patients before and 1-3 months after the procedure with their effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* - Older than 18-year-old
* Clincal, radiological (Grade 3-4) and laboratory examinations ara related with diagnosis of hip joint osteoarthirtis
* Despite of previous medical and physical treatment, VAS score > 5 and above
* Norological examination without critical motor and sensory deficency
* Patients who sign informed consent.

Exclusion Criteria:

* Coagulation disorders (bleeding diathesis)
* Usage of antitrombotic, anticoagulant medications
* Sepsis and local infection on intervention area
* Allergic to any of drugs which is used in intervention
* Without informed consent approval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale comparison | Baseline
  VAS is the most common pain scale. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Visual Analog Scale comparison | 1.month
  VAS is the most common pain scale. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Visual Analog Scale comparison | 3.month
  VAS is the most common pain scale. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Halil Cetingok, Ass. Prof, Study Director — Istanbul University
Locations (1):
- Halil Cetingok, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No